CLINICAL TRIAL: NCT02902809
Title: A 52-Week, Open-Label, Multicentre Study to Evaluate the Safety of Tralokinumab in Japanese Adults and Adolescents With Asthma Inadequately Controlled on Inhaled Corticosteroid Plus Long-Acting β2-Agonist
Brief Title: A Study to Evaluate the Safety of Tralokinumab in Adults and Adolescents With Uncontrolled Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to the discontinuation of the tralokinumab asthma program (as per the results of the Phase III study [D2210C00008])
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2210C00029
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Inadequately Controlled Asthma
Keywords: open-label study; tralokinumab; subcutaneous; inadequately controlled asthma; asthma; medium to high-dose of inhaled corticosteroid; long-acting β2-agonist
MeSH Terms: conditions — Asthma | interventions — tralokinumab

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label study to evaluate safety (Experimental): A fixed 300 mg dose every 2 weeks (Q2W) of tralokinumab administered subcutaneously in subjects with inadequately controlled asthma on medium to high-dose of inhaled corticosteroid plus long-acting β2-agonist.
  Interventions: Biological: Tralokinumab open-label

INTERVENTIONS:
Biological: Tralokinumab open-label — Subcutaneous injection; fixed dose; 300 mg
  Other Names: Tralokinumab

SUMMARY:
A 52-Week, Open-Label, Multicentre Study to Evaluate the Safety of Tralokinumab in Japanese Adults and Adolescents with Asthma Inadequately Controlled on Inhaled Corticosteroid plus Long-Acting β2-Agonist

DETAILED DESCRIPTION:
This is a 52-week, open-label, multi-centre study designed to evaluate the safety of tralokinumab in a fixed 300 mg dose every 2 weeks, administered subcutaneously in adults and adolescents with indequately controlled asthma on medium to high dose inhaled corticosteroid plus long acting β-2 antagonist. Approximately 26 Japanese subjects will be recruited to receive 22 completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 - 75 yrs
2. Documented physician-diagnosed asthma
3. Documented treatment with inhaled corticosteroid (ICS) at a total daily dose corresponding to ≥500 µg fluticasone propionate dry powder formulation equivalents and a long-acting beta-2 agonist (LABA)
4. Pre-bronchodilator (BD) forced expiratory volume at one second (FEV1) value of ≥40% of their Predicted Normal Value (PNV)
5. Asthma Control Questionnaire-6 (ACQ-6) score ≥1.5

Exclusion Criteria:

1. Pulmonary disease other than asthma
2. History of anaphylaxis following any biologic therapy
3. Hepatitis B, C or HIV
4. Pregnant of breastfeeding
5. History or cancer
6. Current tobacco smoking or a history or tobacco smoking for ≥10 pack-years
7. Previous receipt of tralokinumab

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kaneko, MD, PhD, Principal Investigator — Yokohama City University Graduate School of Medicine
Locations (3):
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Itabashi-ku
  - Research Site, Yokohama

REFERENCES:
- [Derived] Panettieri RA Jr, Wang M, Braddock M, Bowen K, Colice G. Tralokinumab for the treatment of severe, uncontrolled asthma: the ATMOSPHERE clinical development program. Immunotherapy. 2018 Mar 1;10(6):473-490. doi: 10.2217/imt-2017-0191. Epub 2018 Mar 14. PMID 29536781
- See also: Statistical Analysis Plan — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4175&filename=D2210C00029_Statistical%20Analysis%20Plan-ed-2_16Feb2018_redacted05Apr2019_Redacted_val.pdf
- See also: Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4175&filename=d2210c00029-csp-v2_15June2017_redacted05April2019_Redacted_val.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with asthma inadequately controlled on inhaled corticosteroid plus long-acting beta 2 agonist were recruited at 4 sites in Japan from 01 November 2016 until study termination on 24 January 2018. No adolescent participants were enrolled in the study.
Pre-assignment Details: Of all enrolled participants, 3 were considered screen failures and 28 participants were received study treatment. Following initial screening, there was a run-in period of up to 2 weeks to allow adequate time for eligibility criteria to be evaluated prior to entry to planned 52-week treatment period followed by a 14 week extended follow-up period.
Groups:
- Tralokinumab 300 mg Every 2 Weeks (Q2W): Participants were administered with tralokinumab 300 milligram (mg) subcutaneous injection every 2 weeks for 52 weeks.
Period: Overall Study
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
Started | 28
Treatment Received | 28
Treatment Completed | 2
Completed | 0
Not Completed | 28
Not completed — Discontinuation of asthma program | 28

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants enrolled and who received at least 1 dose of investigational product irrespective of their protocol adherence and continued participation in the study.
Groups:
- Tralokinumab 300 mg Every 2 Weeks (Q2W): Participants were administered with tralokinumab 300 mg subcutaneous injection every 2 weeks for 52 weeks.
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was development of an undesirable medical condition or deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to product. An undesirable medical condition can be symptoms, signs or the abnormal results of an investigation. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including run-in or washout periods, even if no study treatment has been administered. A SAE was an AE occurred during any study phase that fulfils one or more of the following criteria: death; immediately life-threatening, in-patient or prolongation of existing hospitalization; persistent or significant disability/incapacity or substantial disruption of ability to conduct normal life functions; congenital abnormality or birth defect; important medical event that may jeopardise participant or may require medical intervention to prevent one of the outcomes listed above.
Time Frame: From Screening (Day -14) up to 14 weeks after end of treatment (Week 66).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
Number analyzed (Participants) | 28
Participants
  Any AE | 21
  Any AE with outcome of death | 0
  Any SAE (including events with outcome of death) | 1
  Any AE leading to discontinuation of study drug | 1

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Blood and urine samples for determination of clinical chemistry, haematology and urinalysis parameters were taken at the times. Changes in haematology and clinical chemistry variables between baseline and each subsequent scheduled assessment were evaluated. Baseline is defined as the last available value measured prior to the first dose of study treatment. The change from baseline is defined as the treatment period value minus the baseline period value. Absolute values were compared to the relevant reference range and classified as low (below range), normal (within range or on limits) or high (above range). The AstraZeneca extended reference ranges were used for laboratory variables (where they exist). All values (absolute and change) falling outside the reference ranges were flagged. Urinalysis data were categorised as negative (0), trace or positive (+) at each time point.
Time Frame: From Screening (Day -14) up to 14 weeks after end of treatment (Week 66).
Population: No participants were analysed as the study was terminated due to discontinuation of tralokinumab asthma program. Study was reported in a synopsis format. Individual listings of clinical laboratory parameters were evaluated for safety signal.
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Abnormal Physical Examinations
Description: Physical examination included assessment of general appearance, skin, head and neck (including eyes, ears, nose, mouth and throat), lymph nodes, abdomen, musculoskeletal (including spine and extremities), cardiovascular, respiratory, and neurological systems. Criteria for abnormal physical findings were based on investigator's discretion.
Time Frame: From Screening (Day -14) up to 14 weeks after end of treatment (Week 66).
Population: The study was terminated due to discontinuation of tralokinumab asthma program. Study was reported in a synopsis format. Individual listings were evaluated for safety signal. Any new finding(s) or aggravated existing finding(s), judged as clinically significant by the Investigator, were reported as an AE.
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Vital signs that were planned to be assessed included parameters such as pulse, systolic blood pressure, diastolic blood pressure, respiration rate and body temperature.
Time Frame: From Screening (Day -14) up to 14 weeks after end of treatment (Week 66).
Population: The study was terminated due to discontinuation of tralokinumab asthma program. Study was reported in a synopsis format. Individual listings were evaluated for safety signal. No summary table was developed.
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Participants With 12-Lead Electrocardiogram (ECG) Abnormalities
Description: The ECG assessments were performed using an ECG device prior to blood drawing, spirometry, investigational product administration and bronchodilator administration. ECG data and evaluation was planned to be performed by the site Investigator.
Time Frame: At Day -14 and Week 52.
Population: as for outcome 4
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Screening (Day -14) to study termination (Approximately 60 weeks).
Description: The safety analysis set included all participants enrolled and who received at least 1 dose of investigational product irrespective of their protocol adherence and continued participation in the study.
Arm/Group | Tralokinumab 300 mg Every 2 Weeks (Q2W)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab 300 mg Every 2 Weeks (Q2W) (N=28)
Chronic tonsillitis (Infections and infestations) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab 300 mg Every 2 Weeks (Q2W) (N=28)
Viral upper respiratory tract infection (Infections and infestations) | 10 (20)
Influenza (Infections and infestations) | 4 (4)
Oral herpes (Infections and infestations) | 2 (3)
Acute sinusitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (4)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Sciatica (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Hyperaemia (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Injection site reaction (General disorders) | 9 (57)
Asthenia (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (3)
Thirst (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was terminated due to discontinuation of tralokinumab asthma program. Study was reported in a synopsis format. Individual listings of laboratory variables, physical examinations, vitals and ECG were evaluated for safety signal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02902809/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT02902809/SAP_001.pdf